CLINICAL TRIAL: NCT06570863
Title: To Evaluate the Effects of Systemic Probiotics (Lactobacillus), Antibiotics (Doxycycline 100mg) and Local Application of Metronidazole Gel (25%) As an Adjuvant to Non-surgical Periodontal Therapy
Brief Title: To Evaluate the Effects of Systemic Probiotics & Antibiotics and Local Application of Antibiotics As an Adjuvant to NSPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr fizza khalid (Other)
Responsible Party: Sponsor-Investigator, Dr fizza khalid, Dr Fizza khalid, Assistant Professor. principal investigator, Baqai Medical University
Organization: Baqai Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BaqaiMU
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Periodontitis; Adult
Keywords: periodontitis; probiotics; antibiotics; local application
MeSH Terms: conditions — Periodontitis | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1: Scaling and root Planning (SRD) + Antibiotics (Experimental): doxycycline 100 mg 2 stat the first day followed by od for 14 days
  Interventions: Other: Antibiotics(doxycycline)
- Group 2: SRD + Probiotics (Experimental): Probiotic powder of Lactobacillus Reuteri. After mechanical debridement patient will be prescribed with Lactobacillus rhamnosus SP1 [(2x107colony forming units (CFU)/ day)] (Macrofood S.A., Santiago de Chile, Chile) for 1 month. The dose would be one sachet taken orally daily. The sachets presented to the patients would be identical. Individuals will be instructed to dissolve 1 sachet in water (150 mL) and ingest it once a day after brushing their teeth.
  Interventions: Other: Probiotics
- Group 3: SRD + Metronidazole Gel 25% (Experimental): After mechanical debridement, 25% of metronidazole gel was administered into the periodontal pockets. The gel was applied with a parojet syringe provided with a blunt cannula.
  Interventions: Other: Metronidazole gel 25%

INTERVENTIONS:
Other: Antibiotics(doxycycline) — doxycycline 100 mg 2 stat the first day followed by od for 14 days
  Arms: Group 1: Scaling and root Planning (SRD) + Antibiotics
Other: Probiotics — Probiotic powder of Lactobacillus Reuteri. After mechanical debridement patient will be prescribed with Lactobacillus rhamnosus SP1 [(2x107colony forming units (CFU)/ day)] (Macrofood S.A., Santiago de Chile, Chile) for 1 month. The dose would be one sachet taken orally daily. The sachets presented to the patients would be identical. Individuals will be instructed to dissolve 1 sachet in water (150 mL) and ingest it once a day after brushing their teeth.
  Arms: Group 2: SRD + Probiotics
Other: Metronidazole gel 25% — After mechanical debridement, 25% of metronidazole gel was administered into the periodontal pockets. The gel was applied with a parojet syringe provided with a blunt cannula
  Arms: Group 3: SRD + Metronidazole Gel 25%

SUMMARY:
Background:

Periodontitis is defined as "an inflammatory disease of the supporting tissues of the teeth caused by specific microorganisms or groups of specific microorganisms, resulting in progressive destruction of the periodontal ligament and alveolar bone with pocket formation, recession or both. It has been shown that systemic administration of antibiotics results in changes in plaque flora, reduction in gingivitis and decrease in the rate of bone resorption. In systemic administration, however, the drug must be given in high doses in order to maintain effective concentration of the drug in the gingival crevicular fluid. Whereas recent literature supports use of Local antibiotic therapy which involves the direct placement of an antimicrobial agent into sub gingival sites. The primary goal in using an intra-pocket device for the delivery of an antibacterial agent is the achievement and maintenance of therapeutic levels of the drug for the required period of time. More over use of probiotics is increasing in dentistry, Probiotics are bacterial strains usually isolated from human commensal microbiota and adequately characterized for strain identity, content, stability, and proven health effects. They come in food supplements (cheese, yoghurt, milk, lozenges) with microbial elements.

The purpose of this study is to test the clinical effects of systemic antibiotics, local delivery of 25% of metronidazole gel and probiotics after scaling and root planning in periodontitis.

Objective:

To evaluate the effects of Probiotics (Lactobacillus), antibiotics (Doxycycline 100mg) and metronidazole gel (25%) as an adjuvant to non-surgical periodontal therapy on pocket depth, clinical attachment loss and bleeding on probing after one month of intervention among patients with periodontitis.

Methods:

All study participants meeting the inclusion criteria of the study will be allocated to one of the three groups (Group 1= SRP + Antibiotics, Group 2 = SRP + probiotics and Group 3 = SRP+ LDD) through randomization. After the baseline recording of clinical periodontal parameters, non-surgical periodontal therapy will be done and Group A will be given antibiotic therapy for 14 days, group B will be given probiotics for 1 month and group C will be given LDD after NSPT. After 1-month follow-up and recording of all the clinical parameters will be done.

DETAILED DESCRIPTION:
The most common inflammatory condition of soft and hard tissues, Periodontitis is an infection caused by microorganisms results in progressive destruction of the periodontal ligament and alveolar bone with pocket formation and clinical attachment loss (2) The progression of periodontal disease depends on the interaction among the bacterial agent, environment, and host's defence mechanisms (1,2) According to the Global Burden of Disease Study (2016), periodontal disease is the 11th most prevalent condition. It affects about 20% - 50% of the population worldwide (3) involving approximately 743 million individuals. It has been reported that periodontal disease increases with age (4) and owing to improved life expectancy, 70% of the current world population is above 65years of age (4). The frequency of the periodontal diseases in Pakistani population is no exemption. Its prevalence in Punjab is estimated to be 37%, 40% in Sindh, 20% in Khyber Pakhtunkhwa and 3% in Baluchistan. (5) The primary goal for treatment of Periodontitis includes removing of microbial agents and risk factors to prevent progression of disease and establishing a maintained periodontal tissue (6). Non-surgical periodontal therapy includes scaling and root debridement which aims to abolish bacterial plaque and calculus from supra gingival and sub gingival areas and to restore periodontal health. After NSPT a number of topical antiseptics, anti-inflammatory and antibiotics agents are available which promotes healing of periodontal tissues and are beneficial in treatment of Periodontitis. (5,6) Systemic antibiotics enter the periodontal tissues and periodontal pocket via saliva and gingival crevicular fluid and can affect microorganisms which are unapproachable by NSPT. Additionally, systemic antibiotic therapy has the potential to suppress periodontal pathogens residing on the tongue or other oral surfaces, and by this delaying sub gingival recolonization of pathogens. (7,8) The use of systemic antibiotics as a part of the periodontal therapy has been recommended as an adjunctive therapy in specific situations such as with patients showing progressive periodontal breakdown even after conventional mechanical treatment. (8,9) In the last 25 years, reports stating that systemically administered antibiotics are excreted via saliva and gingival fluid, have triggered great interest in antibiotic therapy. (9) It has been shown that systemic administration of antibiotics results in changes in plaque flora, reduction in gingivitis and decrease in the rate of bone resorption. In systemic administration, however, the drug must be given in high doses in order to maintain effective concentration of the drug in the gingival crevicular fluid as the drug passes the blood stream, gingival crevicular fluid and saliva. (9) Akalin et al compared the clinical efficacies of systemic Doxycycline and local Doxycycline (LD) in the treatment of chronic periodontitis in 45 patients and the results showed that the Local Doxycycline treatment provided significantly higher Probing Depth reduction than the Systemic Doxycycline treatment. (10) The various disadvantages of systemic antibiotics had led to the introduction of local drug delivery as the treatment option. It was in the year 1979, Dr. Max Goodson et al first proposed the concept of controlled delivery in the treatment of periodontitis. (11) Local drug delivery involves the direct placement of an antimicrobial agent into sub gingival sites. The primary goal in using an intra-pocket device for the delivery of an antibacterial agent is the achievement and maintenance of therapeutic levels of the drug for the required period. This inhibits or kills the pathogens, without any harm to the tissues. Studies suggest that the critical period of exposure of the pocket to an antibacterial agent is in the range of 7-10 days. (10,12) Noyan et al reported local metronidazole in combination with scaling and root planning to be more effective than systemic metronidazole in terms of producing both clinical and microbial improvements in adult periodontitis patients. (13) Probiotics conventionally used in the field of medicine are also used to regulate and treat periodontal disease by the application of bacterial replacement therapy. Nowadays, probiotics are commonly used in the oral health perspective because of antibiotic resistance and frequent recolonization of treated sites with pathogenic bacteria. (14) Oral probiotics bacteria bind and colonize periodontal tissue including hard non-shedding surfaces and become part of the biofilm. A few studies have shown that probiotics Lactobacillus strains have been effective in reducing gingival inflammation and diminishing P. gingivalis in the saliva and subgingival plaque. Additionally, Lactobacilli have been found to minimize the levels of periodontal pathogens on the tongue which considered as a significant reservoir for their dissemination and thereby, indirectly minimize the colonization of subgingival plaque by periodontal pathogens. (15) The purpose of this study is to evaluate the effects of Probiotics (Lactobacillus), antibiotics (Doxycycline 100mg) and metronidazole gel (25%) as an adjuvant to non-surgical periodontal therapy on pocket depth, clinical attachment loss and bleeding on probing after one month of intervention among patients with periodontitis.

Methodology:

This Randomized Controlled Clinical trial was conducted at the Department of Periodontology Baqai Dental college. Patients visiting OPD for routine procedure were examined for periodontitis.

Sample size calculation, based on a study previously published (Akalin et al.,2003), was made for the primary outcome variable (CAL), considering a standard deviation of 0.58 and a mean difference between the groups of 0.69. According to the calculation, 32 patients were needed in each group to provide 90% power with and α of 0.05. sample size will be increased 10% to overcome dropout. i-e 40 participants in each group.

Out of 160 patients 90 patients had periodontitis and out of those 40 patients met our inclusion criteria and were selected in this trial after signing the consent form. Inclusion included Male/ female, 35-65 years of age with minimal 12 natural teeth excluding 3rd molars, Patients having Periodontitis (Stage 1 or 2 Grade A) (CAL: 3-4mm) and bleeding on probing in more than 20% sites and systematically healthy. Participants excluded from our research were those with systemic or topical use of antibiotic or undergone any surgical or nonsurgical periodontal therapy in past 6 months, any history of allergies, smokers and smokeless tobacco users, pregnant woman and lactating mothers. Patients with periodontitis were explained the research study after signing the consent form all the enrolled participants went through a detailed history. Principal investigator recorded all the clinical parameters bleeding on probing (BoP), pocket depth (PD) and clinical attachment loss (CAL). These parameters were recorded with the help of UNC-15 probe at the baseline (day 0) and 4 weeks from all the teeth excluding 3rd molars. After complete periodontal examination baseline recordings were recorded for bleeding on probing it was measured by placing the UNC 15 probe into the pocket and wait for 30 seconds,0 = No bleeding on probing, 1 = Bleeding on probing. Probing Depth (PD) was measured from gingival margin to base of the pocket using UNC-15 Probe on four sites of each tooth (Mesio-Buccal, Mesio-lingual,Disto-buccal and Disto-lingual). Clinical Attachment Loss (CAL) was measured from cement-o-enamel junction to base of the pocket with UNC-15 probe on each tooth. After this all participants underwent scaling and root debridement (SRD) through both hand and ultrasonic scaler (Woodpacker). After SRD participant according to their allocated groups. All study participants were allocated to one of the three groups (Group A= scaling and root debridement (SRD) + antibiotics, Group B = SRD + probiotics and Group C = SRD+ Local application) through randomization. For randomization sealed opaque envelopes were used. Participants were asked by the appointed research assistant to pick one envelope containing the name of the therapy which was provided to them. Throughout the study period blinding was maintained (participant were blinded and outcome assessor was blinded in the study) with the help of research assistant who held all the details related to the study groups and treatment strategy till the completion of the trial and complete analysis of the research data. All participants were guided to perform brushing technique (modified bass technique) and instructed to use similar toothpaste (Colgate) during study period, twice daily.

Interventions:

Group 1: Scaling and root Planning (SRD) + Antibiotics doxycycline 100 mg 2 stat the first day followed by od for 14 days. Group 2: SRD + Probiotics Probiotic powder of Lactobacillus Reuteri. After mechanical debridement patient will be prescribed with Lactobacillus rhamnosus SP1 [(2x107colony forming units (CFU)/ day)] (Macrofood S.A., Santiago de Chile, Chile) for 1 month. The dose would be one sachet taken orally daily. The sachets presented to the patients would be identical. Individuals will be instructed to dissolve 1 sachet in water (150 mL) and ingest it once a day after brushing their teeth.

Group 3: SRD + Metronidazole Gel 25% After mechanical debridement, 25% of metronidazole gel was administered into the periodontal pockets. The gel was applied with a parojet syringe provided with a blunt cannula.

After 4 weeks all clinical parameters will be recorded again. (Primary outcome PD, CAL, BOP)

ELIGIBILITY:
Inclusion Criteria:

1. Male/ female, 35-65 years of age.
2. Minimum 12 natural teeth excluding 3rd molars.
3. Patients having Periodontitis (Stage 1 or 2 Grade A) (CAL: 3-4mm).
4. Bleeding on probing in more than 20% sites.
5. Systematically healthy.

Exclusion Criteria:

1. Systemic or topical use of antibiotic.
2. undergone any surgical or nonsurgical periodontal therapy in past 6 months. history of allergies.
3. smokers and smokeless tobacco users.
4. pregnant woman and lactating mothers.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
CAL | 1 month
  clinical attachment loss
PD | 1 month
  pocket deapth
BOP | 1 month
  bleeding on probing

CONTACTS AND LOCATIONS:
Locations (1):
- Baqai Medical University, Karachi, Sindh, Pakistan